CLINICAL TRIAL: NCT03125746
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles and the Antitumor Activity of LXI-15029 Alone or in Combination With Exemestane at Single Ascending Dose and Multiple Ascending Doses in Chinese Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of LXI-15029 in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OE861501
Record Dates: First submitted 2017-03-31; First posted 2017-04-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LXI-15029 (Experimental)
  Interventions: Drug: LXI-15029
- LXI-15029+Exemestane (Experimental)
  Interventions: Drug: LXI-15029+Exemestane

INTERVENTIONS:
Drug: LXI-15029 — The investigational product for this study is LXI-15029 capsule, which can be administered orally and the specification included 10 mg and 50 mg. There will be about 6 cohorts during the monotherapy period. LXI-15029 capsules will be administered in a therapeutic cycle of 28 days twice a day orally. The patients will be given LXI-15029 continuously, in a therapeutic cycle of 28 days. Patients will continue therapy with LXI-15029 if good safety and tolerability were assessed by investigators after 1 cycle treatment. The treatment will continue until progression or occurrence of unmanageable toxicity.
  Arms: LXI-15029
Drug: LXI-15029+Exemestane — The combined drug in the combined therapy period of this study (investigational product) is Exemestane tablet (specification 25 mg). Exemestane should be taken at similar time every day in case of multiple doses (Cycle 1 Day 1 to Cycl 1 Day 28). If one dose was missed (e.g., forgetting, vomiting, etc.), this dose could not be made up and should be administered at next scheduled time point. And the dose of LXI-15029 will be determinated by safety review committee after dose escalation
  Arms: LXI-15029+Exemestane

SUMMARY:
1. To evaluate the safety and tolerability of LXI-15029 in Chinese patients with advanced malignant solid tumors in monotherapy period, including confirmation of the maximum tolerated dose (MTD) of monotherapy. 2.To evaluate the safety and tolerability of LXI-15029 in Chinese postmenopausal patients with metastatic or locally advanced breast cancer with estrogen receptor (+) and human epidermal growth factor receptor 2 (-) in combined with Exemestane period , including confirmation of the maximum tolerated dose(MTD) of the combined therapy with Exemestane.

ELIGIBILITY:
Inclusion Criteria:

* Monotherapy Period

  1. Patients with signed written informed consent form;
  2. Chinese man or woman, aged 18 to 65 years old;
  3. Patient with histologically or cytologically confirmed, advanced solid tumor after failure of standard of care or without standard of care;
  4. Patients must have at least one measurable lesion as defined by RECIST v1.1 (during dose escalation phase,no measurable lesion as defined by RECIST v1.1 but evaluable lesion could also been enrolled);
  5. Expected survival no less than 12 weeks;
  6. Eastern Cooperative Oncology Group (USA) Performance Status 0 to 1;
  7. Patient of childbearing potential (regardless of man or woman) who is willing to take contraceptive measures from signature of the informed consent form to 3 months after the last dose of investigational product. Negative serum pregnancy test within 7 days prior to the planned first dose of investigational product for female patient of childbearing potential;
  8. Have the ability to communicate with study staff, understand and comply with all the study requirements;
* Combined with Exemestane period

  1. Patients with signed written informed consent form;
  2. Chinese patients aged postmenopausal women to 65 years old;
  3. Postmenopausal patient;
  4. Histologically or cytologically confirmed metastatic or locally advanced breast cancer that is not suitable for surgery or radiotherapy;
  5. Estrogen receptor (+), defined as tumor cells with estrogen receptor (+) ≥1% in immunohistochemistry;
  6. HER2-negative (Human epithelial growth factor receptor 2-negative) tumor;
  7. Measurable lesions in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
  8. Expected survival no less than 12 weeks;
  9. Eastern Cooperative Oncology Group (USA) Performance Status 0 to 1;
  10. Have the ability to communicate with study staff, understand and comply with all the study requirements;

Exclusion Criteria:

* Monotherapy Period:

  1. Previous antitumor therapy or any surgical operation within 4 weeks prior to administration of the first dose of study drug;
  2. Treatment with myeloid hematopoietic growth factor within 2 weeks prior to use of investigational product;
  3. Patients receiving corticosteroids or immunosuppressive agents within 4 weeks prior to administration of the first dose of study drug;
  4. Use of potent-to-moderate cytochrome metabolism enzyme CYP3A4 inhibitor and inducer prior to treatment or during washout period;
  5. Known allergy to LXI-15029 or similar products (mammalian target of rapamycin (mTOR) inhibitor or dual mTOR inhibitor) or other components of LXI-15029;
  6. Previous or receiving of PI3K or mTOR inhibitors (e.g., BKM120, everolimus, AZD8055 or AZD2014, etc.);
  7. History, symptoms or signs of spinal compression, brain metastasis or meningeal metastasis, or manifestations of edema or progression in radiology;
  8. History of other tumors within 5 years, except cured carcinoma in situ of cervix or cutaneous basal cell carcinoma;
  9. The toxicity induced by treatment unable to be recovered or stabilized to grade 1 or below except alopecia (common terminology criteria on adverse event version 4.03 (CTCAE 4.03));
  10. Hemotology and coagulation abnormal defined in protocol;
  11. Hepatic function abnormal defined in protocol;
  12. Renal function abnormal defined in protocol;
  13. Cholesterol > 300 mg/dl or 7.75 mmol/L, and/or triglyceride > 2.5 × ULN;
  14. Previous history of type 1 or 2 diabetes, or abnormal fasting blood glucose >126 mg/dL(>7 mmol/L) at screening;
  15. Cardiovascular system diseases;
  16. Patients with active upper peptic ulcer, refractory nausea and vomiting, or other conditions that were known to affect absorption, distribution, metabolism or elimination of drugs;
  17. Patients with chronic obstructive emphysema, pulmonary fibrosis or pneumonia that could significantly affect pulmonary function at discretion of the investigator;
  18. Infectious Diseases defined in protocol;
  19. Judged by the investigator, any other serious or uncontrolled acute or chronic disease, or laboratory abnormality (including but not limited to cardiovascular, hepatic and renal, as well as neuromuscular system), and alcohol consumption, drug abuse that could possibly increase the risk for study or interfere with study conduction and result analysis;
  20. Pregnant or lactating women;
  21. Previous enrollment in this study or participation in this investigational therapy;
  22. Participation in other clinical study during the last 30 days prior to Visit 1
  23. At discretion of the Investigator, the patient is unsuitable for participation in this study for any reasons;
  24. Patient of poor compliance.
* Combined with Exemestane period

  1. Previous antitumor therapy or any surgical operation within 4 weeks prior to administration of the first dose of study drug;
  2. Treatment with myeloid hematopoietic growth factor within two weeks prior to use of investigational product;
  3. Patients receiving corticosteroids or immunosuppressive agents within 4 weeks prior to administration of the first dose of study drug;
  4. Use of potent-to-moderate cytochrome metabolism enzyme CYP3A4 inhibitor and inducer prior to treatment or during washout period
  5. Previous use of Exemestane tablet;
  6. Known allergy to LXI-15029 or similar products (mTOR inhibitor or dual mTOR inhibitor) or other component of LXI-15029;
  7. Previous or receiving of PI3K or mTOR inhibitors (e.g., BKM120, everolimus, AZD8055 or AZD2014, etc.;
  8. Visceral crisis of breast cancer, not suitable for endocrine therapy;
  9. Inflammatory breast cancer;
  10. History, symptoms or signs of spinal compression, brain metastasis or meningeal metastasis, or manifestations of edema or progression in radiology;
  11. History of other tumors within 5 years, except cured carcinoma in situ of cervix or cutaneous basal cell carcinoma;

      Exclusion criteria on concomitant disease and organ function:
  12. The toxicity induced by treatment unable to be recovered or stabilized to grade 1 or below except alopecia (CTCAE 4.03);
  13. Hemotology and coagulation abnormal defined in protocol;
  14. Hepatic function abnormal defined in protocol;
  15. Renal function abnormal defined in protocol;
  16. Cholesterol > 300 mg/dl or 7.75 mmol/L, and/or triglyceride > 2.5 × ULN;
  17. Previous history of type 1 or 2 diabetes, or abnormal fasting blood glucose >126 mg/dL(>7 mmol/L) at screening;
  18. Cardiovascular system abnormal defined in protocol;
  19. Patients with active upper peptic ulcer, refractory nausea and vomiting, or other conditions that were known to affect absorption, distribution, metabolism or elimination of drugs;
  20. Patients with chronic obstructive emphysema, pulmonary fibrosis or pneumonia that could significantly affect pulmonary function at discretion of the investigator;
  21. Infectious Diseases defined in protocol;
  22. Judged by the investigator, any other serious or uncontrolled acute or chronic disease, or laboratory abnormality, and alcohol consumption, drug abuse that could possibly increase the risk for study or interfere with study conduction and result analysis;
  23. Previous enrollment in this study or participation in this investigational therapy;
  24. Participation in other clinical study during the last 30 days prior to Visit 1
  25. At discretion of the Investigator, the patient is unsuitable for participation in this study for any reasons;
  26. Patient of poor compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2021-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | When subject complete 1 cycle (28 days) treatment with safety and tolerability assessment by investigators.
  To evaluate the safety and tolerability of LXI-15029 through evaluation of the incidence and severity of adverse event (Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE, 4.03))

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) | When subject complete 1 cycle (28 days) treatment
  Characterising the pharmacokinetics (PK) profile of LXI-15029
Area Under the Curve (AUC) | When subject complete 1 cycle (28 days) treatment
  Characterising the pharmacokinetics (PK) profile of LXI-15029
Tmax | When subject complete 1 cycle (28 days) treatment
  Characterising the pharmacokinetics (PK) profile of LXI-15029

OTHER OUTCOMES:
Best objective response | Estimated to be up to 6 months
  Best Objective Response per Response Evaluation Criteria in Solid Tumours Criteria (RECIST) 1.1 for target and non target lesions assessed by CT, MRI or X-ray; Complete Response (CR), Disappearance of all target lesions since baseline; Partial Response (PR), At least a 30 percent decrease in the sum of diameters of target lesions; Progressive Disease (PD), At least a 20 percent increase in the sum of diameters of target lesions and an absolute increase of at least 5mm
Progression-free survival (PFS) | Estimated to be up to 6 months
  Duration from treatment start to the time of disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Wang J, Gui L, Mu Y, Wang J, Chi Y, Liu Z, Li Q, Xu B. Phase I dose escalation study and pilot efficacy analysis of LXI-15029, a novel mTOR dual inhibitor, in Chinese subjects with advanced malignant solid tumors. BMC Cancer. 2023 Dec 6;23(1):1200. doi: 10.1186/s12885-023-11578-8. PMID 38057772
- [Derived] Zhang Q, Zhang Y, Chen Y, Qian J, Zhang X, Yu K. A Novel mTORC1/2 Inhibitor (MTI-31) Inhibits Tumor Growth, Epithelial-Mesenchymal Transition, Metastases, and Improves Antitumor Immunity in Preclinical Models of Lung Cancer. Clin Cancer Res. 2019 Jun 15;25(12):3630-3642. doi: 10.1158/1078-0432.CCR-18-2548. Epub 2019 Feb 22. PMID 30796032